CLINICAL TRIAL: NCT01727960
Title: The Effect of Education on Decreasing the Prevalence and Severity of Neck and Shoulder Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Sun Young Park, Doctor, Soonchunhyang University Hospital
Other Study IDs: EduNSP
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Korean; Male; Adolescents
Keywords: Education; Neck pain; Shoulder pain; Prevalence; Associated factors; Students
MeSH Terms: conditions — Neck Pain; Shoulder Pain | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Korean Male Adolescents: students from two academic high schools
  Interventions: Behavioral: Education and posture correction

INTERVENTIONS:
Behavioral: Education and posture correction — a lecture concerning the fine posture for health and exercises

SUMMARY:
Neck and shoulder pain (NSP) is fairly common among high school students in Korea. Presumably, the high prevalence of NSP in Korean adolescents is a consequence of an inappropriate static position for a prolonged period of time. We suspect that proper education and posture correction for Korean adolescents may decrease the prevalence or severity of NSP. Although several studies have focused on the etiology of NSP during adolescence, few studies have addressed the management or prevention of NSP in adolescents, despite its high prevalence in this age group. The aims of this prospective study was to identify the effects of education, in terms of recognition of this issue and posture correction, on prevalence and severity of NSP in Korean adolescents

ELIGIBILITY:
Inclusion Criteria:

* high school students

Exclusion Criteria:

* deny to participate

Ages: 16 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: students from two academic high schools in the city of Seoul 912 students ranging in age from participated.
Sampling Method: Non-Probability Sample
Enrollment: 1302 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
NRS score of neck and shoulder pain | 3 months later
  numeric rating scale (NRS; range, 0-100)of neck and shoulder pain during the 1-week period preceding follow-up

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | 3 months later
  Total NDI scores were interpreted as follows: 0-4, no disability; 5-14, mild disability; 15-24, moderate disability; 25-34, severe disability; >34, complete disability

CONTACTS AND LOCATIONS:
Locations (1):
- Soonchunhyang Univsrsity Hospital, Seoul, South Korea